CLINICAL TRIAL: NCT03665285
Title: A Phase 1/2, Open-Label, Dose-Escalation, Safety and Tolerability Study of NC318 in Subjects With Advanced or Metastatic Solid Tumors
Brief Title: A Safety and Tolerability Study of NC318 in Subjects With Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NextCure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NC318-01
Record Dates: First submitted 2018-09-06; First posted 2018-09-11 (Actual); Results first posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Advanced or Metastatic Solid Tumors; Lung Cancer; Breast Cancer; Head and Neck Squamous Cell Carcinoma; Endometrial Cancer; Melanoma; CRC; Urothelial Carcinoma; Cholangiocarcinoma
Keywords: Advanced Cancer; Metastatic Cancer; NC318; Immunotherapy; PD-L1; Dose Escalation; Biomarker; PK; Cohort Expansion; Solid Tumor
MeSH Terms: conditions — Lung Neoplasms; Breast Neoplasms; Squamous Cell Carcinoma of Head and Neck; Endometrial Neoplasms; Melanoma; Carcinoma, Transitional Cell; Cholangiocarcinoma; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Phase 1 will utilize a 3 + 3 design to explore escalating dose levels. Phase 2 Dose Expansion will further evaluate the safety, tolerability, preliminary efficacy, and PK/PD activity of NC318 at the RP2D utilizing a Simon 2-stage design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- NC318 8mg (Experimental): Phase 1 Dose Escalation (Cohort -1): Subjects received NC318 IV at 8mg Q2W until disease progression, withdraw of consent, or intolerable toxicity (whichever comes first).
  Interventions: Drug: NC318
- NC318 24mg (Experimental): Phase 1 Dose Escalation (Cohort 1): Subjects received NC318 IV at 24mg Q2W until disease progression, withdraw of consent, or intolerable toxicity (whichever comes first).
  Interventions: Drug: NC318
- NC318 80mg (Experimental): Phase 1 Dose Escalation/Safety Expansion (Cohort 2): Subjects received NC318 IV at 80mg Q2W until disease progression, withdraw of consent, or intolerable toxicity (whichever comes first).
  Interventions: Drug: NC318
- NC318 240mg (Experimental): Phase 1 Dose Escalation/Safety Expansion (Cohort 3): Subjects received NC318 IV at 240mg Q2W until disease progression, withdraw of consent, or intolerable toxicity (whichever comes first).
  Interventions: Drug: NC318
- NC318 400mg (Experimental): Phase 1 Dose Escalation/Safety Expansion (Cohort 4): Subjects received NC318 IV at 400mg Q2W until disease progression, withdraw of consent, or intolerable toxicity (whichever comes first).
  Interventions: Drug: NC318
- NC318 800mg (Experimental): Phase 1 Dose Escalation (Cohort 5): Subjects received NC318 IV at 800mg Q2W until disease progression, withdraw of consent, or intolerable toxicity (whichever comes first).
  Interventions: Drug: NC318
- NC318 1600mg (Experimental): Phase 1 Dose Escalation (Cohort 6): Subjects received NC318 IV at 1600mg Q2W until disease progression, withdraw of consent, or intolerable toxicity (whichever comes first).
  Interventions: Drug: NC318
- Dose Expansion: 400mg Q2W (Experimental): Phase 2 Dose Expansion (400mg): Subjects received NC318 IV at 400mg Q2W until disease progression, withdraw of consent, or intolerable toxicity (whichever comes first).
  Interventions: Drug: NC318
- Dose Expansion: 800mg QW (Experimental): Phase 2 Dose Expansion (800mg): Subjects received NC318 IV at 800mg QW for 8 weeks, then Q2W thereafter until disease progression, withdraw of consent, or intolerable toxicity (whichever comes first).
  Interventions: Drug: NC318

INTERVENTIONS:
Drug: NC318 — NC318 is an experimental antibody drug that may make the immune response more active against cancer.

SUMMARY:
This research study is studying a new drug, NC318, as a possible treatment for advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 or older.
* Willingness to provide written informed consent for the study.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1.
* Subjects with advanced unresectable and/or metastatic solid tumors.
* Subjects who have disease progression after treatment with available therapies that are known to confer clinical benefit, or who are intolerant to treatment, or who refuse standard treatment. Note: There is no limit to the number of prior treatment regimens.
* Presence of measurable disease based on RECIST v1.1. Tumor lesions situated in a previously irradiated area, or in an area subjected to other locoregional therapy, are not considered measurable unless there has been demonstrated progression in the lesion.
* Able to provide pretreatment tumor tissue sample at Screening.
* Subjects of childbearing potential (defined as female subjects who have not undergone surgical sterilization with a hysterectomy and/or bilateral oophorectomy and are not postmenopausal, defined as ≥ 12 months of amenorrhea not caused by reversible conditions, diseases, or medications) and non-sterilized male subjects must agree to take appropriate precautions to avoid pregnancy or fathering children (with at least 99% certainty) from screening through 90 days after the last dose of study drug.

Exclusion Criteria:

* Inability to comprehend or unwilling to sign the Informed Consent Form.
* Screening laboratory values of:

  1. Absolute neutrophil count < 1.5 × 10^9/L
  2. Platelets < 100 × 10^9/L
  3. Hemoglobin < 9 g/dL or < 5.6 mmol/L
  4. Serum creatinine > 1.5 × institutional upper limit of normal (ULN)
  5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) > 2.5 × ULN
  6. Total bilirubin > 1.5 × ULN.
  7. International normalized ratio (INR) or prothrombin time (PT) > 1.5 × ULN or activated partial thromboplastin time (aPTT) > 1.5 × ULN
* Transfusion of blood products (including platelets or red blood cells) or administration of colony-stimulating factors (including granulocyte colony-stimulating factor, granulocyte macrophage colony-stimulating factor, or recombinant erythropoietin) within 7 days before the first administration of study drug.
* Receipt of anticancer medications or investigational drugs within the following intervals before the first administration of study drug:

  1. ≤ 14 days for chemotherapy, targeted small molecule therapy, or radiation therapy. Subjects must also not require chronic use of corticosteroids and must not have had radiation pneumonitis because of a treatment. A 1-week washout is permitted for palliative radiation to non-central nervous system (CNS) disease with medical monitor approval. Note: Bisphosphonates and denosumab are permitted medications.
  2. ≤ 28 days for prior immunotherapy or persistence of active cellular therapy (e.g., chimeric antigen receptor T cell therapy; other cellular therapies must be discussed with the medical monitor to determine eligibility).
  3. ≤ 28 days for a prior monoclonal antibody used for anticancer therapy except for denosumab.
  4. ≤ 7 days for immune-suppressive-based treatment for any reason. Note: Use of inhaled or topical steroids or corticosteroid use for radiographic procedures is permitted. Note: The use of corticosteroids equivalent to prednisone </= 10mg/day is allowed.
  5. ≤ 28 days or 5 half-lives (whichever is longer) before the first dose for all other investigational study drugs or devices.
  6. ≤ 14 days for COVID-19 vaccine.
* Has not recovered to ≤ Grade 1 from toxic effects of prior therapy (including prior immunotherapy) and/or complications from prior surgical intervention before starting therapy.
* Receipt of a live vaccine within 30 days of planned start of study therapy.
* Active autoimmune disease that required systemic treatment in the past (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs).
* Known active CNS metastases and/or carcinomatous meningitis.
* Known additional malignancy that is progressing or requires active treatment, or history of other malignancy within 2 years of study entry after treatment with curative intent.
* Has a history of (non-infectious) pneumonitis / interstitial lung disease that required steroids or has current pneumonitis / interstitial lung disease.
* Documented known activating or driver mutations (i.e. EGFR mutations/amplification, BRAF mutations, ALK alterations, etc.) which have not been previously treated with a standard of care targeted therapy.
* Subjects with screening QTc interval >470 milliseconds are excluded.
* Uncontrolled systemic fungal, bacterial, viral, or other infection despite appropriate anti-infection treatment.
* Evidence of hepatitis B virus (HBV) or hepatitis C virus (HCV), unless the hepatitis is considered to be cured.
* Known history of HIV (HIV 1 or HIV 2 antibodies).
* Known allergy or reaction to any component of study drug or formulation components.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 90 days after the last dose of study treatment.
* Any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of study drug and attending required study visits; pose a significant risk to the subject; or interfere with interpretation of study data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Han Myint, MD, Study Director — NextCure, Inc.
Locations (6):
- United States (6):
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - Yale University Cancer Center, New Haven, Connecticut
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Laura and Isaac Perlmutter Cancer Center, New York, New York
  - Pennsylvania Cancer Specialists and Research Institute, Gettysburg, Pennsylvania
  - NEXT Oncology, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 109 participants took part in the study at 6 investigative sites in the United States from 01 October 2018 to 11 April 2023.
Pre-assignment Details: The dose-escalation consisted of 7 planned cohorts (NC318 IV doses of 8 mg to 1600 mg). Phase 1b was a safety expansion of 3 cohorts (80 mg, 240 mg, and 400 mg). 49 participants were enrolled in Phase 1. A RP2D of 400 mg Q2W was initially evaluated in Phase 2 (N=47); an alternative RP2D of 800 mg weekly for 8 cycles, followed by 800 mg Q2W thereafter (N=13) was also evaluated.
Period: Overall Study
Arm/Group | NC318 8mg | NC318 24mg | NC318 80mg | NC318 240mg | NC318 400mg | NC318 800mg | NC318 1600mg | Dose Expansion: 400mg Q2W | Dose Expansion: 800mg QW
Started | 4 | 4 | 10 | 12 | 11 | 4 | 4 | 47 | 13
Completed | 3 | 3 | 5 | 7 | 9 | 3 | 2 | 19 | 11
Not Completed | 1 | 1 | 5 | 5 | 2 | 1 | 2 | 28 | 2
Not completed — Started New Anticancer Treatment | 1 | 1 | 2 | 4 | 1 | 1 | 2 | 15 | 1
Not completed — Disease Progression | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 7 | 1
Not completed — Hospice | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) includes all subjects enrolled in the study who received at least one full dose of NC318.
Groups:
- Total: Total of all reporting groups
Arm/Group | NC318 8mg | NC318 24mg | NC318 80mg | NC318 240mg | NC318 400mg | NC318 800mg | NC318 1600mg | Dose Expansion: 400mg Q2W | Dose Expansion: 800mg QW | Total
Number analyzed (Participants) | 4 | 4 | 10 | 12 | 11 | 4 | 4 | 47 | 13 | 109
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 4 | 7 | 8 | 3 | 3 | 23 | 5 | 58
  >=65 years | 1 | 2 | 6 | 5 | 3 | 1 | 1 | 24 | 8 | 51
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 6 | 7 | 6 | 3 | 2 | 30 | 7 | 65
  Male | 2 | 2 | 4 | 5 | 5 | 1 | 2 | 17 | 6 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 3 | 3 | 0 | 0 | 5 | 2 | 15
  Not Hispanic or Latino | 3 | 4 | 9 | 9 | 8 | 4 | 4 | 41 | 10 | 92
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 6 | 1 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
  White | 4 | 4 | 10 | 9 | 9 | 4 | 4 | 35 | 7 | 86
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 5 | 3 | 12
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 10 | 12 | 11 | 4 | 4 | 47 | 13 | 109

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events as Assessed by CTCAE v5.0
Description: The number of participants who have had at least one TEAE during the study.
Time Frame: From enrollment through up to 90 days after end of treatment, an average of 1 year
Population: The Safety Analysis Set (SAS) will include all the subjects who receive any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | NC318 8mg | NC318 24mg | NC318 80mg | NC318 240mg | NC318 400mg | NC318 800mg | NC318 1600mg | Dose Expansion: 400mg Q2W | Dose Expansion: 800mg QW
Number analyzed (Participants) | 4 | 4 | 10 | 12 | 11 | 4 | 4 | 47 | 13
Participants | 4 | 4 | 10 | 12 | 11 | 4 | 4 | 45 | 12

2. Secondary Outcome: Objective Response Rate (ORR) as Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Description: To assess antitumor activity/efficacy by evaluating objective response rate (ORR), defined as the percentage of participants who experienced a complete response (CR; disappearance of all target lesions) or a partial response (PR; at least a 30% decrease in the sum of diameters of target lesions) based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Time Frame: Approximately 1 year
Population: The full analysis set (FAS) includes all subjects enrolled in the study who received at least one full dose of NC318.
Measure: Count of Participants; unit: Participants
Arm/Group | NC318 8mg | NC318 24mg | NC318 80mg | NC318 240mg | NC318 400mg | NC318 800mg | NC318 1600mg | Dose Expansion: 400mg Q2W | Dose Expansion: 800mg QW
Number analyzed (Participants) | 4 | 4 | 10 | 12 | 11 | 4 | 4 | 47 | 13
Participants | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0

3. Secondary Outcome: Duration of Response (DoR) as Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Description: To assess antitumor activity/efficacy by evaluating duration of response (DoR), defined as the time from the first documented complete response or partial response per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 to the first documented progressive disease or death due to any cause, whichever occurs first. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: Approximately 1 year
Population: The full analysis set (FAS) includes all subjects enrolled in the study who received at least one full dose of NC318.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NC318 8mg | NC318 24mg | NC318 80mg | NC318 240mg | NC318 400mg | NC318 800mg | NC318 1600mg | Dose Expansion: 400mg Q2W | Dose Expansion: 800mg QW
Number analyzed (Participants) | 4 | 4 | 10 | 12 | 11 | 4 | 4 | 47 | 13
months | NA [NA to NA] — Insufficient number of participants with events. | NA [NA to NA] — Insufficient number of participants with events. | NA [NA to NA] — Insufficient number of participants with events. | NA [NA to NA] — Insufficient number of participants with events. | NA [NA to NA] — Insufficient number of participants with events. | NA [NA to NA] — Insufficient number of participants with events. | NA [NA to NA] — Insufficient number of participants with events. | 8.11 [NA to NA] — Insufficient number of participants with events. | NA [NA to NA] — Insufficient number of participants with events.

4. Secondary Outcome: Disease Control Rate (DCR) as Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Description: To assess antitumor activity/efficacy by evaluating disease control rate (DCR), defined as the proportion of participants in whom a documented complete response, partial response, or stable disease is observed as the best overall response per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Time Frame: Approximately 1 year
Population: The full analysis set (FAS) includes all subjects enrolled in the study who received at least one full dose of NC318.
Measure: Count of Participants; unit: Participants
Arm/Group | NC318 8mg | NC318 24mg | NC318 80mg | NC318 240mg | NC318 400mg | NC318 800mg | NC318 1600mg | Dose Expansion: 400mg Q2W | Dose Expansion: 800mg QW
Number analyzed (Participants) | 4 | 4 | 10 | 12 | 11 | 4 | 4 | 47 | 13
Participants | 3 | 0 | 8 | 2 | 5 | 3 | 2 | 14 | 1

5. Secondary Outcome: Progression-free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Description: To evaluate progression-free survival (PFS), defined as the time from the first dose of NC318 to the first occurrence of documented progressive disease or death due to any cause, whichever occurs first. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Approximately 1 year
Population: The full analysis set (FAS) includes all subjects enrolled in the study who received at least one full dose of NC318.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NC318 8mg | NC318 24mg | NC318 80mg | NC318 240mg | NC318 400mg | NC318 800mg | NC318 1600mg | Dose Expansion: 400mg Q2W | Dose Expansion: 800mg QW
Number analyzed (Participants) | 4 | 4 | 10 | 12 | 11 | 4 | 4 | 47 | 13
months | NA [2.82 to NA] — The median and upper limit of the confidence interval were not estimable due to limited number of participants with events. | 1.32 [0.97 to NA] — The upper limit of the confidence interval was not estimable due to limited number of participants with events. | 5.72 [1.47 to 10] | 1.86 [1.1 to NA] — The upper limit of the confidence interval was not estimable due to limited number of participants with events. | 2.54 [1.82 to 5.14] | 3.93 [1.79 to NA] — The upper limit of the confidence interval was not estimable due to limited number of participants with events. | 3.29 [0.54 to NA] — The upper limit of the confidence interval was not estimable due to limited number of participants with events. | 2.04 [1.82 to 2.25] | 1.79 [0.79 to 1.97]

6. Secondary Outcome: Overall Survival (OS)
Description: To evaluate overall survival (OS), defined as the time from the first dose of NC318 to death due to any cause.
Time Frame: Approximately 1 year
Population: The full analysis set (FAS) includes all subjects enrolled in the study who received at least one full dose of NC318.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NC318 8mg | NC318 24mg | NC318 80mg | NC318 240mg | NC318 400mg | NC318 800mg | NC318 1600mg | Dose Expansion: 400mg Q2W | Dose Expansion: 800mg QW
Number analyzed (Participants) | 4 | 4 | 10 | 12 | 11 | 4 | 4 | 47 | 13
months | NA [NA to NA] — The median and confidence intervals were not estimable due to limited number of participants with event. | NA [1.71 to NA] — The median and upper limit of the confidence interval were not estimable due to limited number of participants with event. | NA [NA to NA] — The median and confidence intervals were not estimable due to limited number of participants with event. | 11.04 [1.54 to NA] — The upper limit of the confidence interval was not estimable due to limited number of participants with event. | 6.18 [3.25 to NA] — The upper limit of the confidence interval was not estimable due to limited number of participants with event. | NA [4.07 to NA] — The median and upper limit of the confidence interval were not estimable due to limited number of participants with event. | NA [1.28 to NA] — The median and upper limit of the confidence interval were not estimable due to limited number of participants with event. | NA [NA to NA] — The median and confidence intervals were not estimable due to limited number of participants with event. | 3.55 [0.95 to NA] — The upper limit of the confidence interval was not estimable due to limited number of participants with event.

7. Secondary Outcome: Maximum Plasma Concentration (Cmax) of NC318
Description: To evaluate the Maximum Plasma Concentration (Cmax) of NC318
Time Frame: Days 1, 2, and 3 of Cycles 1 and 5 and Day 1 of Cycles 2, 3, 6, 9, 13, 17, and 21. Each cycle is 7 days during Cycles 1-8 and 14 days thereafter.
Population: The PK analysis set (PAS) will include all the subjects whose blood samples are collected for PK analysis. PK analysis only took place during the dose escalation portion of the study.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | NC318 8mg | NC318 24mg | NC318 80mg | NC318 240mg | NC318 400mg | NC318 800mg | NC318 1600mg
Number analyzed (Participants) | 4 | 4 | 10 | 12 | 11 | 4 | 4
ng/mL | 3010 (2194) | 5020 (774) | 17130 (5120) | 55025 (12393) | 97816 (19174) | 352500 (310095) | 329750 (99399)

8. Secondary Outcome: Area Under the Curve (AUC) of NC318
Description: To evaluate the Area Under the Curve (AUC) of NC318
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | NC318 8mg | NC318 24mg | NC318 80mg | NC318 240mg | NC318 400mg | NC318 800mg | NC318 1600mg
Number analyzed (Participants) | 4 | 4 | 10 | 12 | 11 | 4 | 4
h*ng/mL | 171933 (NA) — SD was below the lower limit of detection. | 112327 (NA) — SD was below the lower limit of detection. | 290486 (115984) | 724225 (538755) | 1324013 (688403) | 4335767 (2288217) | 9837043 (5163985)

9. Secondary Outcome: Half-life (t1/2) of NC318
Description: To evaluate the half-life (t1/2) of NC318
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | NC318 8mg | NC318 24mg | NC318 80mg | NC318 240mg | NC318 400mg | NC318 800mg | NC318 1600mg
Number analyzed (Participants) | 4 | 4 | 10 | 12 | 11 | 4 | 4
hours | 46.16 (NA) — SD was below lower limit of detection. | 24.62 (NA) — SD was below lower limit of detection. | 46.41 (10.68) | 34.81 (13.15) | 32.25 (10.37) | 32.67 (6.57) | 32.71 (6.0)

ADVERSE EVENTS:
Time Frame: From enrollment through up to 90 days after end of treatment, an average of 1 year
Description: The severity of AEs will be assessed using NCI CTCAE v5.0 Grades 1 through 4. The NCI CTCAE v5.0 severity of Grade 5 will not be used; AEs resulting in death will be graded accordingly using Grades 1 through 4 and have the outcome noted as fatal.
Arm/Group | NC318 8mg | NC318 24mg | NC318 80mg | NC318 240mg | NC318 400mg | NC318 800mg | NC318 1600mg | Dose Expansion: 400mg Q2W | Dose Expansion: 800mg QW
All-Cause Mortality (participants affected / at risk) | 0/4 | 2/4 | 0/10 | 4/12 | 3/11 | 1/4 | 1/4 | 7/47 | 6/13
Serious Adverse Events (participants affected / at risk) | 2/4 | 3/4 | 4/10 | 8/12 | 4/11 | 1/4 | 3/4 | 16/47 | 5/13
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 10/10 | 12/12 | 10/11 | 4/4 | 4/4 | 42/47 | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NC318 8mg (N=4) | NC318 24mg (N=4) | NC318 80mg (N=10) | NC318 240mg (N=12) | NC318 400mg (N=11) | NC318 800mg (N=4) | NC318 1600mg (N=4) | Dose Expansion: 400mg Q2W (N=47) | Dose Expansion: 800mg QW (N=13)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Death nos (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Disease Progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 2 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Endometrial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Encephalitis autoimmune (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Device occlusion (Product Issues) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pelvic Pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NC318 8mg (N=4) | NC318 24mg (N=4) | NC318 80mg (N=10) | NC318 240mg (N=12) | NC318 400mg (N=11) | NC318 800mg (N=4) | NC318 1600mg (N=4) | Dose Expansion: 400mg Q2W (N=47) | Dose Expansion: 800mg QW (N=13)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 3 | 3 | 4 | 1 | 1 | 6 | 4
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Diplopia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Extraocular muscle paresis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 2 | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 2 | 2 | 3 | 0 | 0 | 6 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Abdominal pain UPPER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 4 | 3 | 1 | 0 | 1 | 4 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 4 | 3 | 2 | 1 | 0 | 3 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 4 | 3 | 3 | 1 | 1 | 8 | 3
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 3 | 0 | 0 | 1 | 9 | 4
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 1 | 1 | 3 | 1 | 0 | 6 | 1
Face oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 4 | 2 | 1 | 1 | 1 | 12 | 2
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0
Oedema peripheral (General disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 4 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 1 | 3 | 1 | 1 | 0 | 3 | 1
Supraclavicular fossa pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chorioretinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 7 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 1
Amylase increased (Investigations) | 0 | 0 | 2 | 1 | 2 | 0 | 1 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 2 | 1 | 1 | 1 | 4 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 3 | 2 | 1 | 1 | 1 | 2
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 2
Blood calcium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 2
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 2
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 2 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 7 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 2 | 0 | 1 | 1 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 2 | 2 | 1 | 1 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2 | 2 | 1 | 2 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 3 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2 | 3 | 2 | 1 | 3 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 5 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 4 | 1
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Burning sensation (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 3 | 1 | 0 | 0 | 0 | 5 | 1
Dysaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fine motor skill dysfunction (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 2 | 0 | 1 | 1 | 0 | 2 | 4 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 4 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 8 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 4 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 4 | 0 | 2 | 1 | 1 | 5 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Extremity necrosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Peripheral embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI cannot publish study results before the first multi-center publication. If a multi-center publication is not submitted within 12 months after the end of the study at all sites, or if Sponsor confirms there will be no multi-center publication, the PI may publish study results. However, PI will allow Sponsor at least 30 days to review any publication of study results and Sponsor may request an additional 60 days to review the publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-03): https://cdn.clinicaltrials.gov/large-docs/85/NCT03665285/Prot_SAP_000.pdf